CLINICAL TRIAL: NCT00907179
Title: Pemetrexed and LBH589 in Previously-Treated Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Pemetrexed and LBH589 in Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Widespread use firstline Pemetrexed; slow recruitment; funding withdrawn..
Sponsor: University of Pittsburgh (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-036
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Panobinostat; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalation (Experimental): Phase I: Determine the highest and safest dosage of LBH589 (15 mg, 20 mg, and 30 mg). If the 15 mg dosage causes too many side effects, a back-up dosage of 10 mg will be used instead of the 15 mg.
  Pemetrexed 500mg/m2 IV, day 1, every 21 days, on the first day of the week LBH589 is given
  Interventions: Drug: LBH 589; Drug: Pemetrexed

INTERVENTIONS:
Drug: LBH 589 — LBH589 three-times-a-week (doses will be at least 2 days apart, e.g. Monday, Wednesday, Friday), until disease progression or intolerable toxicities LBH589 will start the week prior to the first pemetrexed cycle and PD studies will be performed (week -1).
  Dose level: 1 LBH589: 10 mg Pemetrexed: 500 mg/m2
  Dose level: 2 LBH589: 15 mg Pemetrexed: 500 mg/m2
  Dose level: 3 LBH589: 20 mg Pemetrexed: 500 mg/m2
  Dose level: 4 LBH589: 30 mg Pemetrexed: 500 mg/m2
  Other Names: Panobinstat
Drug: Pemetrexed — Pemetrexed 500mg/m2 IV, day 1, every 21 days, on the first day of the week LBH589 is given.
  Other Names: Alimta

SUMMARY:
LBH589 is a drug that may slow down the growth of cancer cells or kill cancer cells by blocking certain enzymes. LBH589 has shown effects against cancer in laboratory studies and in studies using animals; however, it is not known if this medicine will show the same activity in humans. As of May 2006, approximately 100 patients have received treatment with either an intravenous or capsule form of LBH589. Only the capsule form of LBH589 will be used in this study. In addition, information from other research studies and laboratory studies suggests that this study drug may help to treat lung cancer.

The main goal during the Phase I portion of this research study is to find out the highest and safest dose of LBH589 that can be given in combination with pemetrexed in subjects with lung cancer without causing severe side effects. The main goal of the Phase II portion of this study is to find how the patient's lung cancer responds to the LBH589 in combination with pemetrexed.

This study will also investigate how the patient's body processes the combination of LBH589 and pemetrexed. To determine this, the investigators will measure the amount of study drug in the patient's blood. This will be done with a series of blood tests, called pharmacokinetic (PK) tests. Other purposes of this study will be to determine the side effects of LBH589 in combination with pemetrexed and whether or not this combination is effective in treating your type of cancer.

DETAILED DESCRIPTION:
Objectives

1. To determine the maximum tolerated dose of LBH589 given on a three times weekly schedule when combined with pemetrexed for the treatment of patients with advanced thoracic malignancies, except squamous cell carcinoma of the lung (phase I part).
2. To determine the overall response rate and non-progression rate (clinical benefit rate) and progression-free survival of the combination of LBH589 and pemetrexed in patients with previously-treated advanced NSCLC (phase II part).
3. To determine the pharmacodynamic effects of LBH589 and pemetrexed on levels of histone deacetylase (HDAC) 1 and 6 in peripheral blood mononuclear cells, as well as on levels of vascular endothelial growth factor (VEGF) levels in the blood.
4. To identify biomarkers in baseline, archival tumor tissue that may correlate with antitumor efficacy.

Subject population Phase I: We will enroll patients treated with any number of prior regimen and all thoracic malignancies, except squamous cell carcinoma of the lung.

Phase II: We will enroll patients with recurrent or progressive NSCLC who have received 1 prior chemotherapy regimen (1 additional regimen in the setting of initial curative treatment is allowed if completed >1 year earlier).

Treatment plan

* Pemetrexed 500mg/m2 IV, day 1, every 21 days, on the first day of the week LBH589 is given.
* LBH589 three-times-a-week (doses will be at least 2 days apart, e.g. Monday, Wednesday, Friday), until disease progression or intolerable toxicities LBH589 will start the week prior to the first pemetrexed cycle and pharmacodynamic (PD) studies will be performed (week -1)

Study design and sample size:

This is a phase I/II study. Phase I: 9-18 patients (estimated); Phase II: 17-41 patients (estimated).

ELIGIBILITY:
Inclusion Criteria:

1. Phase I only: any number of prior regimens is allowed and all thoracic malignancies, except squamous cell carcinoma of the lung.
2. Phase II only: Patients with recurrent or progressive advanced stage non-squamous cell NSCLC (no small cell lung cancer/SCLC component) who have received 1 prior chemotherapy regimen for advanced NSCLC. Chemotherapy as part of initially potentially curative therapy that was completed <1 year counts as 1 prior regimen. Prior erlotinib or one other biologic regimen is also allowed.
3. Measurable disease (RECIST) (for phase II part only)
4. Patients may not have received prior pemetrexed or histone deacetylase inhibitor (HDACi) therapy, including valproic acid, for the treatment of any medical condition.
5. ECOG (Eastern Cooperative Oncology Group) Performance Status of ≤ 2
6. Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
7. Patients must meet the following laboratory criteria:

   * Hematology:

     * Absolute neutrophil count (ANC) ≥ 1500/mm³
     * Platelets ≥ 100,000/mm³
     * Hemoglobin ≥ 9 g/dL
   * Biochemistry:

     * Total Bilirubin within normal institutional limits.
     * Aspartate aminotransferase/glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/glutamic pyruvic transaminase (ALT/SGPT) ≤ 2.5 x upper limit of normal (ULN)
     * Creatinine clearance 45 ml/min or higher calculated using the Cockcroft-Gault formula
   * Total serum calcium (corrected for serum albumin) or ionized calcium within normal limits (WNL)
   * Serum potassium ≥ WNL
   * Serum sodium ≥ WNL
   * Serum albumin ≥ WNL
   * Patients with any elevated Alkaline Phosphatase due to bone metastasis can be enrolled
8. Baseline multiple uptake gated acquisition scan (MUGA) or ECHO must demonstrate left ventricular ejection fraction (LVEF) ≥ the lower limit of the institutional normal.
9. Thytoid stimulating hormone (TSH) and free T4 within normal limits (patients may be on thyroid hormone replacement)
10. Blood pressure of <140/90.
11. Patients must have fully recovered from the effects of any prior surgery, chemotherapy or radiation therapy. A minimum time period of 3 weeks should elapse between the completion of extensive radiation therapy for recurrent/metastatic disease and enrollment in the study. A minimum of 4 weeks should elapse between the completion of chemotherapy or any experimental therapy and enrollment in the study. At least 2 weeks should have elapsed from prior erlotinib or other biologic therapy.
12. If patient has history of brain metastases, brain lesions should have been treated with surgery and/or radiation and be stable on repeat imaging.
13. No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, unless there is a 3- year disease-free interval.
14. Patients should temporary stop certain Nonsteroidal Anti-inflammatory Drug (NSAIDS) starting 5 days prior to protocol therapy, as described in 6.5.1.
15. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment and must be willing to use two methods of contraception one of them being a barrier method or abstain from sexual activity during the study and for 3 months after last study drug administration. Sexually active males and their female partners must agree to use two methods of accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study.
16. All patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

1. Prior HDAC, deacetylase (DAC), HSP90 inhibitors or valproic acid for the treatment of cancer
2. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
3. Impaired cardiac function including any one of the following:

   * Screening ECG with a QTc > 450 msec confirmed by central laboratory prior to enrollment to the study
   * Patients with congenital long QT syndrome
   * History of sustained ventricular tachycardia
   * Any history of ventricular fibrillation or torsades de pointes
   * Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible.
   * Patients with a myocardial infarction or unstable angina within 6 months of study entry
   * Congestive heart failure (NY Heart Association class III or IV)
   * Right bundle branch block and left anterior hemiblock (bifascicular block)
4. Uncontrolled hypertension. Patients with history of hypertension must be well-controlled (≤150/100) on a stable regimen of anti-hypertensive therapy.
5. Concomitant use of drugs with a risk of causing torsades de pointes (See Appendix 1.-1)
6. Concomitant use of Cytochrome (CYP3A4) inhibitors (See Appendix 1-2) is not allowed. The use of cytochrome (CYP2D6) substrates (Appendix 1, table 0-3) should be done with caution. If drugs that are CYP2D6 substrates arte to be continued, patients should be carefully monitored and may require dose titration or dose reduction of the CYP2D6 substrate.
7. Patients with unresolved diarrhea > CTCAE (NCI common terminology criteria for adverse events ) grade 1
8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
9. Other concurrent severe and/or uncontrolled medical conditions
10. Patients who have received chemotherapy, any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
11. Concomitant use of any anti-cancer therapy or radiation therapy.
12. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589.
13. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom
14. Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
15. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
16. Patients with squamous cell carcinomas will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of LBH589 given on a three times weekly schedule when combined with pemetrexed for the treatment of patients with advanced thoracic malignancies, except squamous cell carcinoma of the lung (phase I part) | 6 months

SECONDARY OUTCOMES:
Determine the overall response rate and non-progression rate (clinical benefit rate) and progression-free survival of the combination of LBH589 and pemetrexed in patients with previously-treated advanced NSCLC (phase II part). | 1 year
Determine the pharmacodynamic effects of LBH589 and pemetrexed on levels of HDAC 1 and 6 in peripheral blood mononuclear cells, as well as on levels of VEGF levels in the blood. | 1 year
Identify biomarkers in baseline, archival tumor tissue that may correlate with antitumor efficacy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States